CLINICAL TRIAL: NCT06361303
Title: The Happiest Baby, Inc. SNOO Postmarket Surveillance Study
Status: Recruiting | Type: Observational
Sponsor: Happiest Baby, Inc. (Industry)
Responsible Party: Principal Investigator, Christopher Laine, Principal Research Scientist, Happiest Baby, Inc.
Other Study IDs: PS230001; PS230001 / PSS001 (Other: US FDA)
Record Dates: First submitted 2024-04-03; First posted 2024-04-11 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Infant Death; Serious Injury
MeSH Terms: conditions — Infant Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes | US Export: No

GROUPS / COHORTS (1):
- SNOO users: Caregivers who use the SNOO Bassinet with their infant and who meet eligibility criteria
  Interventions: Device: SNOO Bassinet

INTERVENTIONS:
Device: SNOO Bassinet — This is a non-interventional, prospective observational and descriptive active surveillance study of a cohort of individuals who have purchased or rented a SNOO for use with their infant.

SUMMARY:
This postmarket surveillance study will evaluate the safety of the SNOO Smart Sleeper Bassinet when used for infants who are at high risk for Sudden Unexpected Infant Death (SUID). This study will survey 1000 caregivers of high-risk infants to examine the frequency of death or serious injury occurring in the SNOO Bassinet.

DETAILED DESCRIPTION:
Synopsis:

This postmarket surveillance study will evaluate the ongoing safety of the Happiest Baby, Inc. SNOO Smart Sleeper in accordance with the order issued under Section 522 of the Federal Food, Drug, and Cosmetic Act, issued March 30, 2023

The study will measure rates of adverse events occurring in the SNOO bassinet from a prospectively screened cohort of 1000 infants determined to be at high risk for SUID. The primary endpoints quantify device-related serious injury and/or device-related death. The secondary endpoints include an analysis of SNOO usage patterns in the enrolled population, including infant age during SNOO use, duration of SNOO use, and weaning rationale.

Procedures:

Prospective participants who have purchased or rented SNOO during the study enrollment period will be invited to participate in an electronic eligibility screening survey 1-month after their purchase/rental ship date. Eligible participants will subsequently be invited to participate in a 6-month follow up survey (7 months after their purchase/rental ship date, 6 months post-enrollment) soliciting self-reported outcomes for the study endpoints. The screening and survey questionnaires will be conducted electronically via Qualtrics using a link provided by email, and which may be completed on a smart phone, tablet, or computer.

As enrolled eligible participants complete their final surveys, responses indicating the occurrence of adverse events will be investigated, classified according to severity and device-relatedness, documented, and reported. A final clinical evaluation of the observed SUID rate will be conducted, and will include reference to demographically-matched population statistics pulled from the CDC WONDER database. A full characterization of adverse events and any demographic or usage-related correlates will be reported to the FDA as part of this investigation.

ELIGIBILITY:
Inclusion Criteria:

Infant/caregiver dyads meeting the following inclusion criteria will be eligible for study enrollment:

* Respondent must identify as a primary caregiver of the infant.
* Purchase or rental of SNOO shipped to a U.S. residence during the defined enrollment period.
* Caregivers must be English speakers ages 18 or older residing in the United States.
* Infants must use SNOO during the intended use period (i.e., birth to 6 months).
* Infants must meet at least one of the following criteria for high risk for SUID:

  * Infant race: Black or African American; and/or American Indian or Alaskan Native
  * Maternal education: 12 years or less
  * Low birth weight: <5 pounds 8 ounces (<2500 grams)
  * Last menstrual cycle (LMP) or obstetrical estimate (OE) Gestational age at time of birth: <37 weeks (preterm)
  * Maternal age at time of birth: <25 years
  * Smoking status: Any self-reported maternal smoking during pregnancy

Exclusion Criteria:

* Not primary caregiver
* Does not speak English
* Is not a US resident
* Is not 18 years old or older
* Infant did not use SNOO during the intended use period (i.e., birth to 6 months).
* Infants does NOT meet at least one of the below risk criteria:

  * Infant race: Black or African American; and/or American Indian or Alaskan Native
  * Maternal education: 12 years or less
  * Low birth weight: <5 pounds 8 ounces (<2500 grams)
  * LMP or OE Gestational age at time of birth: <37 weeks (preterm)
  * Maternal age at time of birth: <25 years
  * Smoking status: Any self-reported maternal smoking during pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregivers of infants who use SNOO and are at high risk of SUID, as determined by our eligibility criteria. No more than 25% of enrolled subjects will consist of infant users who exclusively used SNOO from birth to 1 month of age. The majority of enrolled subjects (>50%) will have engaged in SNOO use at some point between 1 and 4 months of infant age. If these enrollment targets are not met, additional subjects will be enrolled until the proposed age distribution and usage criteria are met.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Serious Injury | when infant was 0-6 months old (and still using SNOO)
  Any instance of SNOO-related serious injury reported (Number and percent), with 'serious' defined as 1) life -threatening, 2) Resulting in permanent impairment of body function or permanent damage to body structure, or 3) Necessitates medical or surgical intervention to preclude permanent impairment of a body function or permanent damage to a body structure.
Infant death | when infant was 0-6 months old (and still using SNOO)
  Any instance of device-related infant death (number and percent).

SECONDARY OUTCOMES:
Infant age during SNOO use | when infant was 0-6 months old (and still using SNOO)
  infant age at start and end of SNOO use
Degree of SNOO use | when infant was 0-6 months old (and still using SNOO)
  Frequency of SNOO use [All of the time (>90%); Most of the time (50-90%); Some of the time (10%-49%); None of the time (<10%)]
Weaning rationale | when infant was 0-6 months old (and still using SNOO)
  Reason for ending SNOO use

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Laine, PhD, Principal Investigator — Happiest Baby, Inc.
Locations (1):
- Happiest Baby, Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA site for study — https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfPMA/pss.cfm?t_id=383&c_id=7362